CLINICAL TRIAL: NCT01584193
Title: Ultrasound-guided Subclavian Vein Puncture Versus Cephalic Vein Dissection for Totally Implantable Venous Access Port Implementation: a Single-center Controlled Randomized Superiority Trial
Brief Title: Ultrasound-guided Subclavian Vein Puncture Versus Cephalic Vein Dissection for Venous Access Port Implantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical reasons (institutional reorganization of ambulatory surgery)
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, Professor, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHV 46/11
Record Dates: First submitted 2012-04-21; First posted 2012-04-24 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Vascular Surgical Procedures
Keywords: central venous access port; ultrasound-guided venous puncture; suclavian vein; cephalic vein
MeSH Terms: interventions — Venous Cutdown

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- US-guided subclavian vein puncture (Experimental)
  Interventions: Procedure: Ultrasound-guided subclavian vein puncture
- Cephalic vein dissection (Active Comparator)
  Interventions: Procedure: Cephalic vein dissection

INTERVENTIONS:
Procedure: Ultrasound-guided subclavian vein puncture — Central venous access port implementation through ultrasound-guided subclavian vein puncture and Seldinger technique
  Other Names: US-guided; Seldinger technique
  Arms: US-guided subclavian vein puncture
Procedure: Cephalic vein dissection — Central venous access port implementation through cephalic vein dissection and cutdown
  Other Names: Venous cutdown
  Arms: Cephalic vein dissection

SUMMARY:
The purpose of this study is to compare two different surgical techniques for implementation of totally implantable central venous access ports. Ultrasound-guided suclavian vein puncture is compared to cephalic vein dissection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Informed consent
* Need for central venous access port implementation under local anesthesia

Exclusion Criteria:

* Impaired blood clotting
* Ongoing antiplatelet drugs therapy, except acetylsalicylic acid
* Trauma or surgical past history on both shoulder girdles
* Known central venous thrombosis (subclavian vein, upper vena cava)
* Known pneumothorax
* Septic state
* Agranulocytosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
surgical procedure time | during surgical procedure

SECONDARY OUTCOMES:
primary implementation success rate | during surgical procedure
overall implementation success rate | during surgical procedure
technique conversion rate and causes | during surgical procedure
pain during surgical procedure | during surgical procedure
pain at 5 days | 5 days post-procedure
Pain at 30 days | 30 days post-procedure
Complications rate during surgical procedure | during surgical procedure
  catheter malposition, hemorrhage, hemotoma, hemothorax, pneumothorax
Complications rate at 5 days | 5 days post-procedure
  hematoma, infection, symptomatic venous thrombosis, pneumothorax
Complications rate at 30 days | 30 days post-procedure
  infection, symptomatic venous thrombosis, pneumothorax, venous access port dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Demartines, Study Chair — University Hospital Lausanne, Department of Visceral Surgery
Locations (1):
- University Hospital Lausanne, Department of Visceral Surgery, Lausanne, Canton of Vaud, Switzerland